CLINICAL TRIAL: NCT05021029
Title: The UC Davis Cohort of Pre-Malignant and Malignant GastroIntestinal DisEases (TUMMIE) Study
Brief Title: UC Davis Cohort of Pre-Malignant and Malignant Gastro-Intestinal DisEases Study
Acronym: TUMMIE
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1614453
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Intestinal Metaplasia; Chronic Gastritis; Atrophic Gastritis; Autoimmune Gastritis; Intestinal Dysplasia
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — With patient consents, study team will collect saliva, stool, blood and/or gastric biopsy or gastric juices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To establish a prospective cohort of individuals diagnosed with gastric pre-malignant conditions (chronic gastritis, atrophic gastritis, autoimmune gastritis, intestinal metaplasia, intestinal dysplasia) to monitor and study disease progression. The Investigators will like to survey cohort participants for lifestyle behaviors and environmental exposures associated with gastric pre-malignancy and cancer. Analyzing patient biospecimens to identify and characterize host and microbiome biomarkers associated with initiation and progression of gastric pre-malignancies.

DETAILED DESCRIPTION:
Initially, study coordinators will identify prevalent patients diagnosed with gastric pre-malignancy at UC Davis Health in the last five years or receive a list of eligible patients by a GI doctor at UC Davis Health. These individuals will be sent an invitation letter via mail or by physician, to participate in the study and will be provided with a reply slip authorizing contact by the research team. Individuals willing to participate in the study will be then contacted by research coordinators via phone/mail to:

i) Provide information about the study and answer questions (via phone call, video-conference, letter or email),

ii) Answer study questionnaire

iii) Sign study's informed consent to provide saliva, blood, urine and/or stool samples.

iv) Sign a HIPPA form to obtain permission to retrieve archival tumor blocks and pathology reports

Participants will be also asked for permission to regular re-contact and will be asked to inform study coordinators about future endoscopic appointments, where blood, stomach biopsies and stomach juice samples will be obtained. If the participant agrees, permission will be requested for these samples as well.

To recruit incident participants, the research coordinators will review endoscopic schedules and or be provided a list of patients who fit the criteria to identify participants suspected or diagnosed with gastric pre-malignant diseases. Participants will be asked to consent and asked to fill out a short version survey before their endoscopic procedure. Contact information will be collected (Phone, Address, Email) in order to send the full version of the survey later. Participants will be asked if they would like to donate a blood, saliva and urine sample and will be provided with a stool collection kit for home sampling, which will be returned to the research team in a pre-paid padded envelope. At the appointment, participants will also be asked if they would agree to provide tissue and/or gastric juices that will be obtained by their physician during their procedure or any leftover tissue after histological examination. For specimens requiring histological analyses, only once consents and/or HIPPA waivers are received will any leftover specimens be collected for this research study.

All participants (prevalent and incidence) will be contacted once a year to update surveys, clinical and risk factor information, consent and HIPPA waivers.

Data from the study questionnaire will be analyzed regularly using standard epidemiological methods. Biospecimens will be used for multiple omics approaches and results will be published regularly in medical and scientific journals and conferences.

ELIGIBILITY:
Inclusion Criteria:

1. UCDHS patients
2. Of all races/ethnicities
3. Diagnosed with premalignant conditions such as chronic gastritis, atrophic gastritis, autoimmune gastritis, gastric intestinal metaplasia, gastric intestinal dysplasia or gastic polyps
4. During the last 5 years and current years to come (2015-2025)
5. Some participants may be scheduled for endoscopy

Exclusion Criteria:

* We will not include children (anyone under the age of 18), individuals unable to consent, pregnant women, or prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from University of California Davis Health patients of all races and ethnicities.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Pre-malignant progression | 2024
  Review the number of patients with gastric conditions and any progression to advanced pre-neoplasia/malignancy or cancer and identify and characterize host and microbiome biomarkers associated with initiation and progression of gastric pre-malignancies

SECONDARY OUTCOMES:
Recruitment response rates | 2024
  Review number of patients response rates who donated full/partial biospecimen samples.

CONTACTS AND LOCATIONS:
Overall Officials: Luis G Carvajal-Carmona, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States